CLINICAL TRIAL: NCT01437969
Title: Pharmacogenomics Study on IL28B Genetic Variants in Italian Patients With HCV Chronic Infection naïve to Antiviral Treatment.
Brief Title: Pharmacogenomics Study on IL28B Genetic Variants in Italian Patients With HCV Infection naïve to Treatment.
Status: Completed | Type: Observational
Sponsor: Casa Sollievo della Sofferenza IRCCS (Other)
Collaborators: INMI L Spallanzani IRCCS Roma (Unknown); IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other); Azienda Ospedaliera San Camillo Forlanini (Other); Fondazione IRCCS Policlinico San Matteo di Pavia (Other); Azienda ospedaliera Garibaldi Nesinma Catania (Unknown); Azienda Ospedaliero-Universitaria Careggi (Other); University of Milan (Other); Catholic University, Italy (Other); Ospedale Francesco Ferrari (Other); Ospedale di Canosa di Puglia (Unknown); Ospedale di Venosa (Unknown); Clinica Santa Rita Bari (Unknown); Ospedale SS. Annunziata, Taranto (Unknown); Ospedali Riuniti di Foggia (Other)
Responsible Party: Principal Investigator, Alessandra Mangia, MD, Casa Sollievo della Sofferenza IRCCS
Other Study IDs: EPAT-IL28B
Record Dates: First submitted 2011-09-20; First posted 2011-09-21 (Estimated); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Liver Disease
Keywords: Possible association; between severity; IL28B genetic variants; patients; different HCV genotypes
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA from blood sample

INTERVENTIONS:
Genetic: genotyping and/or sequencing — genotyping and/or sequencing DNA for IL28

SUMMARY:
More than 1.5 millions individuals are infected with HCV in Italy. They are at risk to develop related morbidity and mortality from cirrhosis and hepatocellular carcinoma, unless the evolution of their disease is halted by treatment-induced HCV RNA clearance. Indeed, it is well recognized that a curative antiviral treatment, leading to HCV RNA undetectability 24 weeks after the end of therapy, may prevent the occurrence of complications of HCV chronic liver disease.

Several pre-treatment host and viral factors have been associated with the outcome of pegylated Interferon and Ribavirin treatment. These predictors are relevant as the ability to identify patients with the highest likelihood of achieving HCV RNA clearance may increase the number of patients who agree to be treated and who maintain their adherence to treatment.

Several pre-treatment predictors as HCV genotype, HCV viral load, age, gender, body mass index, stage of fibrosis and race are very well recognized and have been used for many years during the treatment decision-making process. Based on studies of viral kinetics, HCV RNA undetectable at week 4 on treatment has been shown to represent the best on treatment predictor of response. In addition to these well known factors, very recently, a single nucleotide polymorphism (SNP) upstream of the gene IL28B on chromosome 19, coding for IFN-lambda 3 has been identified as associated with both spontaneous and treatment induced HCV RNA clearance.

We have developed the molecular technique needed to evaluate this polymorphism in our laboratory. This technical process was a consequence of the genetics expertise of our research Institute. We have also performed a valuable comparison of the different methods to evaluate this polymorphism. Comparison of different technologies allow us to know the rate of variability between the different assays used.

With this methodology we have evaluated "a posteriori" patients previously enrolled in Randomized Controlled Trial. The results of these studies confirmed the association between IL28B CC allele and a favorable outcome of HCV infection in our geographic area (Mangia et al Gastroenterology 2010; Mangia et al Hepatology 2010, AASLD presentation). We are now interested in prospective evaluation of patients referring to our center at the aim of understanding whether there are differences in the rates of IL28B frequencies in patients with different HCV genotypes.

In fact, we hypothesize that the frequency of IL28B might be different according with different HCV genotypes and that this difference may explain the different rates of response to antiviral treatment reported in patients with HCV infection.

Since we lead a collaborative group of hepatologists named AL-LIVER operating in Puglia, Lazio, Basilicata, Sicilia and Campania regions in Italy we would like to extend this evaluation to our collaborative group to explore in a large number of patients whether the prevalence of CC, CT and TT genotypes is inversely associated with HCV G1, 4, 3 and 2.

DETAILED DESCRIPTION:
This study is a prevalence study involving naïve patients and without links with treatment. Five hundred patients with HCV infection consecutively observed during 2011 will be requested to sign an informed consent at the aim to be tested for genetics. The study will be evaluated and approved by the Central Ethic Committee. It will have a planned duration of 12 months and will involve 15 centers.

All the HCV infected patients previously untreated can be enrolled once they have signed the Informed consent for genetic testing.

Each patient enrolled at the single center will be evaluated for demographical, virological, biochemical, histological and genetic (IL28B) characteristics. In case of unavailable liver biopsy at least APRI score and Fibroscan evaluation should be used to assess the severity of the underlying liver disease. All the blood specimens will be stored and evaluated by a pre-developed TaqMan allelic discrimination assay (Applied Biosystem) or by direct sequencing for IL28B genetic variation. A serum sample will be also stored to evaluate HCV genotype and HCV RNA levels.

Data will be collected in a database that can be used in the future to select patients needing antiviral treatment.

The association between IL28B variants and the other predictors will be explored by means of descriptive statistical analyses. Number of patients, mean, standard deviation, median will be calculated for continuous variables. Absolute frequencies and per cent will be used to describe frequencies parameters

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic HCV infection irrespective of HCV genotype

Exclusion Criteria:

* HCV infected patients previously treated with antiviral drugs; co-infected Patients with HIV or Hepatitis B virus (HBsAg positive)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HCV infected patients previously untreated
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2011-09; Primary Completion 2012-09 (Actual); Study Completion 2022-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Mangia, MD, Principal Investigator — Liver Unit, Casa Sollievo della Sofferenza
Locations (1):
- IRCCS "Casa Sollievo della Sofferenza", San Giovanni Rotondo, Foggia, Italy

REFERENCES:
- [Background] Ge D, Fellay J, Thompson AJ, Simon JS, Shianna KV, Urban TJ, Heinzen EL, Qiu P, Bertelsen AH, Muir AJ, Sulkowski M, McHutchison JG, Goldstein DB. Genetic variation in IL28B predicts hepatitis C treatment-induced viral clearance. Nature. 2009 Sep 17;461(7262):399-401. doi: 10.1038/nature08309. Epub 2009 Aug 16. PMID 19684573
- [Background] Suppiah V, Moldovan M, Ahlenstiel G, Berg T, Weltman M, Abate ML, Bassendine M, Spengler U, Dore GJ, Powell E, Riordan S, Sheridan D, Smedile A, Fragomeli V, Muller T, Bahlo M, Stewart GJ, Booth DR, George J. IL28B is associated with response to chronic hepatitis C interferon-alpha and ribavirin therapy. Nat Genet. 2009 Oct;41(10):1100-4. doi: 10.1038/ng.447. Epub 2009 Sep 13. PMID 19749758
- [Background] Tanaka Y, Nishida N, Sugiyama M, Kurosaki M, Matsuura K, Sakamoto N, Nakagawa M, Korenaga M, Hino K, Hige S, Ito Y, Mita E, Tanaka E, Mochida S, Murawaki Y, Honda M, Sakai A, Hiasa Y, Nishiguchi S, Koike A, Sakaida I, Imamura M, Ito K, Yano K, Masaki N, Sugauchi F, Izumi N, Tokunaga K, Mizokami M. Genome-wide association of IL28B with response to pegylated interferon-alpha and ribavirin therapy for chronic hepatitis C. Nat Genet. 2009 Oct;41(10):1105-9. doi: 10.1038/ng.449. Epub 2009 Sep 13. PMID 19749757
- [Background] Thompson AJ, Muir AJ, Sulkowski MS, Ge D, Fellay J, Shianna KV, Urban T, Afdhal NH, Jacobson IM, Esteban R, Poordad F, Lawitz EJ, McCone J, Shiffman ML, Galler GW, Lee WM, Reindollar R, King JW, Kwo PY, Ghalib RH, Freilich B, Nyberg LM, Zeuzem S, Poynard T, Vock DM, Pieper KS, Patel K, Tillmann HL, Noviello S, Koury K, Pedicone LD, Brass CA, Albrecht JK, Goldstein DB, McHutchison JG. Interleukin-28B polymorphism improves viral kinetics and is the strongest pretreatment predictor of sustained virologic response in genotype 1 hepatitis C virus. Gastroenterology. 2010 Jul;139(1):120-9.e18. doi: 10.1053/j.gastro.2010.04.013. Epub 2010 Apr 24. PMID 20399780
- [Background] Mangia A, Thompson AJ, Santoro R, Piazzolla V, Tillmann HL, Patel K, Shianna KV, Mottola L, Petruzzellis D, Bacca D, Carretta V, Minerva N, Goldstein DB, McHutchison JG. An IL28B polymorphism determines treatment response of hepatitis C virus genotype 2 or 3 patients who do not achieve a rapid virologic response. Gastroenterology. 2010 Sep;139(3):821-7, 827.e1. doi: 10.1053/j.gastro.2010.05.079. Epub 2010 Jun 2. PMID 20621700
- [Background] Afdhal NH, McHutchison JG, Zeuzem S, Mangia A, Pawlotsky JM, Murray JS, Shianna KV, Tanaka Y, Thomas DL, Booth DR, Goldstein DB; Pharmacogenetics and Hepatitis C Meeting Participants. Hepatitis C pharmacogenetics: state of the art in 2010. Hepatology. 2011 Jan;53(1):336-45. doi: 10.1002/hep.24052. PMID 21254181